CLINICAL TRIAL: NCT02756871
Title: Overcoming Perfectionism: A Randomised Controlled Trial of an Online CBT Based Guided Self-help Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14PP31
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2016-04

CONDITIONS: Perfectionism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online guided self-help intervention (Experimental): CBT based online guided self-help intervention. Intervention can be found at www.overcomingperfectionism.co.uk
  Interventions: Other: online guided self-help intervention for perfectionism
- Control (No Intervention): No intervention.

INTERVENTIONS:
Other: online guided self-help intervention for perfectionism — CBT based online guided self-help intervention for perfectionism based on CBT manual for treatment of perfectionism, "Cognitive Behavioural Treatment of Perfectionism" by Sarah Egan, Tracy Wade, Roz Shafran and Martin Antony
  Other Names: Overcoming Perfectionism
  Arms: Online guided self-help intervention

SUMMARY:
The purpose of this study is to assess the effectiveness of CBT based online guided self-help intervention for perfectionism at reducing symptoms of perfectionism and Axis I disorders post-treatment and at six-month follow-up.

DETAILED DESCRIPTION:
Perfectionism is elevated across, and increases risk for a range of Axis I disorders, as well as having a direct negative effect on day to day function. A growing body of evidence shows that cognitive behavioural therapy (CBT) reduces perfectionism and Axis I disorders, with medium to large effect sizes. Given the increased desire for online interventions to facilitate access to evidence-based therapy, web-based CBT self-help interventions for perfectionism have been designed. Existing interventions have not included personalised guidance which has been shown to improve outcome rates.

The purpose of this study is to assess the effectiveness of CBT based online guided self-help intervention for perfectionism at reducing symptoms of perfectionism and Axis I disorders post-treatment and at six-month follow-up.

A randomised controlled trial method is employed, comparing the treatment arm (online guided self-help) with a waiting list control group. Outcomes are examined at three time points, T1 (baseline), T2 (post-intervention at 12 weeks), T3 (follow-up at 24 weeks). Participants will be recruited through universities, online platforms, and social media, and if eligible will be randomised using an online automatic randomiser.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 or over, with no upper age limit.
* Score one standard deviation above published norms on the 'Concern over mistakes' subscale of the Frost Multidimensional Perfectionism Scale (Frost, Marten, Lahart, & Rosenblate, 1990), i.e. a score of ≥ 29 (Flett, Sawatzky, & Hewitt, 1995).
* Be fluent in English.

Exclusion Criteria:

- They report suicidal thoughts or intent prior to commencement of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Frost Multidimensional Perfectionism Scale (Frost et al., 1990) | 6 months
  This self-report measure consists of 36 items grouped into six subscales. Participants respond on a five point scale ranging from 1 = "strongly disagree" to 5 = "strongly agree". The measure has been found to be both reliable and valid for use with non-clinical and clinical populations (Frost et al., 1990; Hewitt & Flett, 1991; Hewitt, Flett, Turnbull-Donovan, & Mikail, 1991). Participants will be considered eligible for inclusion in the study if they score one standard deviation above published norms on the Concern over Mistakes subscale, i.e. a score of ≥ 29. This measure has been amended to reflect participants experience over the past month allowing us to measure change.

SECONDARY OUTCOMES:
Obsessive-Compulsive Inventory - Revised (OCI-R) (Foa et al., 2002) | 6 months
  The OCI-R, a shortened version of the Obsessive-Compulsive Inventory, assesses symptoms of OCD. The measure consists of 18 items (e.g. "I frequently have get nasty thoughts and have difficulty in getting rid of them"). On a five point scale, respondents rate how distressed or bothered they have been in the past month by the symptom described, with responses ranging from "Not at all" to "Extremely." It has been found to have good validity and reliability in both clinical and non-clinical samples (Abramowitz & Deacon, 2006; Foa et al., 2002; Hajcak, Huppert, Simons, & Foa, 2004; Huppert et al., 2007).
Eating Disorder Examination-Questionnaire (EDE-Q) (C. G. Fairburn, 1994) | 6 months
  The EDE-Q assesses for symptoms of the eating disorders: Anorexia Nervosa (AN), Bulimia Nervosa (BN), Binge Eating Disorder (BED) and sub-threshold variants. The measure consists of 28 items rated on a seven point scale appropriate to the item: number of days a symptom has been experienced over the past month, ranging from no days to every day; and for remaining questions (e.g. "How dissatisfied have you been with your weight?") responses ranging from "Not at all" to "Markedly." It has been found to have good reliability, and has been validated for use among clinical and community samples (Aardoom, Dingemans, Op't Landt, & Van Furth, 2012; Carter, Stewart, & Fairburn, 2001; J. M. Mond, Hay, Rodgers, Owen, & Beumont, 2004; Jonathan M Mond et al., 2008; Reas, Grilo, & Masheb, 2006).
Depression, Anxiety and Stress Scales (DASS) (Lovibond & Lovibond, 1996) | 6 months
  The DASS is a 42 item self-report measure of depression, anxiety and stress (e.g. "I found myself getting upset by quite trivial things"), rated on a four point scale ranging from "Did not apply to me at all" to "Applied to me very much or most of the time." It has been shown to be reliable and has been validated for use among clinical and community samples (Brown, Chorpita, Korotitsch, & Barlow, 1997; Crawford & Henry, 2003; Page, Hooke, & Morrison, 2007).
Vancouver Obsessional Compulsive Inventory - Mental Contamination Scale (VOCI-MC) (Radomsky, Rachman, Shafran, Coughtrey, & Barber, 2014) | 6 months
  The VOCI-MC is a self-report measure that assesses symptoms of mental contamination. The measure consists of 20 items (e.g. "Often I look clean but feel dirty), rated on a five point scale ranging from "Not at all" to "Very much." It has been shown to be reliable and valid for use among clinical and community samples (Coughtrey, Shafran, Knibbs, & Rachman, 2012; Coughtrey, Shafran, & Rachman, 2013; Radomsky et al., 2014).
Clinical Perfectionism Questionnaire (CPQ; C. Fairburn et al., 2003a) | 6 months
  This self-report measure consists of 12 items (e.g. "Have you pushed yourself really hard to meet your goals?" and "Have you raised your standards because you thought they were too easy?"). Participants respond on a four point scale ranging from 1 = "not at all" to 4 = "all the time". This measure of clinical perfectionism was created by Fairburn, Cooper and Shafran at the University of Oxford, and has been found to have good reliability and validity in two community samples and an ED sample; participants will be considered eligible for inclusion if they score similarly to this psychiatric population (i.e. a score of ≥ 29) (Egan, Shafran, et al., 2014). This measure has been amended to reflect participants experience over the past week, allowing us to monitor change on a weekly basis.

OTHER OUTCOMES:
Fears of Compassion Scales (FCS; (Paul Gilbert, McEwan, Matos, & Rivis, 2011) | 6 months
  This measure consists of three scales which assess fear of compassion for self (e.g. "I worry that if I start to develop compassion for myself I will become dependent on it"), fear of compassion from others (e.g. "I try to keep my distance from others, even if I know they are kind"), and fear of compassion for others (e.g. "Being too compassionate makes people soft and easy to take advantage of"). The FCS is made up of 38 items in total which are rated on a four point scale ranging from 0 = "Don't agree at all" to 4 = "Completely agree." It has been shown to be reliable, and valid for use among clinical and community samples (P Gilbert et al., 2012; Paul Gilbert et al., 2011).
Rosenberg Self-esteem Scale (Rosenberg, 1965) | 6 months
  This measure of self-esteem consists of 10 items (e.g. "On the whole I am satisfied with myself" and "I wish I could have more respect for myself") and is rated on a four point scale ranging from 1 = "strongly disagree" to 4 = "strongly agree" It has been found to be reliable, and been validated for use among clinical and community samples (Bagley & Mallick, 2001; Ferring & Filipp, 1996; Martín-Albo, Núñez, Navarro, & Grijalvo, 2007; Phillips, Pinto, & Jain, 2004; Schmitt & Allik, 2005; Shaw-Zirt, Popali-Lehane, Chaplin, & Bergman, 2005).
Intolerance of Uncertainty Scale (IoU; (Freeston, Rhéaume, Letarte, Dugas, & Ladouceur, 1994) | 6 months
  The IoU consists of 27 items (e.g. "Uncertainty stops me from having a firm opinion" and "It's unfair not having any guarantees in life"), and is rated on a five point scale ranging from 1 = "Not at all characteristic of me" to 5 = "Entirely characteristic of me." It has been found to be reliable, and has been validated for use among clinical and community samples (Kristine Buhr & Dugas, 2002; Kristin Buhr & Dugas, 2006; Jacoby, Fabricant, Leonard, Riemann, & Abramowitz, 2013).
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS; (Tennant et al., 2007) | 6 months
  The WEMWBS is a 14 item self-report measure of mental well-being that focuses on positive aspects of mental health, including subjective well-being, psychological functioning (including autonomy, competence, self-acceptance, and personal growth), and interpersonal relationships. Examples of items include, "I have been feeling optimistic about the future," "I have been feeling confident," and "I have been dealing with problems well." Participants respond on a five point scale, ranging from 1 = "none of the time" to 5 = "all of the time." The WEMWBS has shown good reliability (0.83) and has been validated for use among student and population samples (Clarke et al., 2011; Maheswaran, Weich, Powell, & Stewart-Brown, 2012; Tennant et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Roz Shafran, PhD, Principal Investigator — UCL Institute of Child Health
Locations (1):
- UCL Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Egan SJ, van Noort E, Chee A, Kane RT, Hoiles KJ, Shafran R, Wade TD. A randomised controlled trial of face to face versus pure online self-help cognitive behavioural treatment for perfectionism. Behav Res Ther. 2014 Dec;63:107-13. doi: 10.1016/j.brat.2014.09.009. Epub 2014 Sep 30. PMID 25461785
- [Result] Aardoom JJ, Dingemans AE, Slof Op't Landt MC, Van Furth EF. Norms and discriminative validity of the Eating Disorder Examination Questionnaire (EDE-Q). Eat Behav. 2012 Dec;13(4):305-9. doi: 10.1016/j.eatbeh.2012.09.002. Epub 2012 Sep 19. PMID 23121779
- [Result] Abramowitz JS, Deacon BJ. Psychometric properties and construct validity of the Obsessive-Compulsive Inventory--Revised: Replication and extension with a clinical sample. J Anxiety Disord. 2006;20(8):1016-35. doi: 10.1016/j.janxdis.2006.03.001. Epub 2006 Apr 18. PMID 16621437
- [Result] Bagley, C., & Mallick, K. (2001). Normative data and mental health construct validity for the Rosenberg Self-Esteem Scale in British Adolescents. International Journal of Adolescence and Youth, 9(2-3), 117-126.
- [Result] Bizeul C, Sadowsky N, Rigaud D. The prognostic value of initial EDI scores in anorexia nervosa patients: a prospective follow-up study of 5--10 years. Eating Disorder Inventory. Eur Psychiatry. 2001 Jun;16(4):232-8. doi: 10.1016/s0924-9338(01)00570-3. PMID 11418274
- [Result] Brown TA, Chorpita BF, Korotitsch W, Barlow DH. Psychometric properties of the Depression Anxiety Stress Scales (DASS) in clinical samples. Behav Res Ther. 1997 Jan;35(1):79-89. doi: 10.1016/s0005-7967(96)00068-x. PMID 9009048
- [Result] Buhr K, Dugas MJ. The Intolerance of Uncertainty Scale: psychometric properties of the English version. Behav Res Ther. 2002 Aug;40(8):931-45. doi: 10.1016/s0005-7967(01)00092-4. PMID 12186356
- [Result] Buhr K, Dugas MJ. Investigating the construct validity of intolerance of uncertainty and its unique relationship with worry. J Anxiety Disord. 2006;20(2):222-36. doi: 10.1016/j.janxdis.2004.12.004. PMID 16464706
- [Result] Carter JC, Stewart DA, Fairburn CG. Eating disorder examination questionnaire: norms for young adolescent girls. Behav Res Ther. 2001 May;39(5):625-32. doi: 10.1016/s0005-7967(00)00033-4. PMID 11341255
- [Result] Clarke A, Friede T, Putz R, Ashdown J, Martin S, Blake A, Adi Y, Parkinson J, Flynn P, Platt S, Stewart-Brown S. Warwick-Edinburgh Mental Well-being Scale (WEMWBS): validated for teenage school students in England and Scotland. A mixed methods assessment. BMC Public Health. 2011 Jun 21;11:487. doi: 10.1186/1471-2458-11-487. PMID 21693055
- [Result] Coughtrey, A. E., Shafran, R., Knibbs, D., & Rachman, S. J. (2012). Mental contamination in obsessive-compulsive disorder. Journal of Obsessive-Compulsive and Related Disorders, 1(4), 244-250.
- [Result] Coughtrey, A. E., Shafran, R., & Rachman, S. (2013). Imagery in mental contamination: A questionnaire study. Journal of Obsessive-Compulsive and Related Disorders, 2(4), 385-390.
- [Result] Crawford JR, Henry JD. The Depression Anxiety Stress Scales (DASS): normative data and latent structure in a large non-clinical sample. Br J Clin Psychol. 2003 Jun;42(Pt 2):111-31. doi: 10.1348/014466503321903544. PMID 12828802
- [Result] Egan SJ, Shafran R, Lee M, Fairburn CG, Cooper Z, Doll HA, Palmer RL, Watson HJ. The Reliability and Validity of the Clinical Perfectionism Questionnaire in Eating Disorder and Community Samples. Behav Cogn Psychother. 2016 Jan;44(1):79-91. doi: 10.1017/S1352465814000629. Epub 2015 Mar 3. PMID 25731214
- [Result] Fairburn, C., Cooper, C., & Shafran, R. (2003a). Clinical Perfectionism Questionnaire. Department of Psychiatry. University of Oxford, United Kingdom.
- [Result] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Result] Ferring, D., & Filipp, S. (1996). Measurement of self-esteem: findings on reliability, validity, and stability of the Rosenberg Scale. Diagnostica, 42(3), 284-292.
- [Result] Foa EB, Huppert JD, Leiberg S, Langner R, Kichic R, Hajcak G, Salkovskis PM. The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess. 2002 Dec;14(4):485-96. PMID 12501574
- [Result] Gilbert P, McEwan K, Matos M, Rivis A. Fears of compassion: development of three self-report measures. Psychol Psychother. 2011 Sep;84(3):239-55. doi: 10.1348/147608310X526511. Epub 2011 Apr 13. PMID 22903867
- [Result] Hajcak G, Huppert JD, Simons RF, Foa EB. Psychometric properties of the OCI-R in a college sample. Behav Res Ther. 2004 Jan;42(1):115-23. doi: 10.1016/j.brat.2003.08.002. PMID 14992204
- [Result] Hewitt, P. L., Flett, G. L., Turnbull-Donovan, W., & Mikail, S. F. (1991). The Multidimensional Perfectionism Scale: Reliability, validity, and psychometric properties in psychiatric samples. Psychological Assessment: A Journal of Consulting and Clinical Psychology, 3(3), 464.
- [Result] Huppert JD, Walther MR, Hajcak G, Yadin E, Foa EB, Simpson HB, Liebowitz MR. The OCI-R: validation of the subscales in a clinical sample. J Anxiety Disord. 2007;21(3):394-406. doi: 10.1016/j.janxdis.2006.05.006. Epub 2006 Jun 30. PMID 16814981
- [Result] Jacoby RJ, Fabricant LE, Leonard RC, Riemann BC, Abramowitz JS. Just to be certain: Confirming the factor structure of the intolerance of uncertainty scale in patients with obsessive-compulsive disorder. J Anxiety Disord. 2013 Jun;27(5):535-42. doi: 10.1016/j.janxdis.2013.07.008. Epub 2013 Aug 6. PMID 23973743
- [Result] Maheswaran H, Weich S, Powell J, Stewart-Brown S. Evaluating the responsiveness of the Warwick Edinburgh Mental Well-Being Scale (WEMWBS): group and individual level analysis. Health Qual Life Outcomes. 2012 Dec 27;10:156. doi: 10.1186/1477-7525-10-156. PMID 23270465
- [Result] Martin-Albo J, Nuniez JL, Navarro JG, Grijalvo F. The Rosenberg Self-Esteem Scale: translation and validation in university students. Span J Psychol. 2007 Nov;10(2):458-67. doi: 10.1017/s1138741600006727. PMID 17992972
- [Result] Mond JM, Hay PJ, Rodgers B, Owen C, Beumont PJ. Validity of the Eating Disorder Examination Questionnaire (EDE-Q) in screening for eating disorders in community samples. Behav Res Ther. 2004 May;42(5):551-67. doi: 10.1016/S0005-7967(03)00161-X. PMID 15033501
- [Result] Mond JM, Myers TC, Crosby RD, Hay PJ, Rodgers B, Morgan JF, Lacey JH, Mitchell JE. Screening for eating disorders in primary care: EDE-Q versus SCOFF. Behav Res Ther. 2008 May;46(5):612-22. doi: 10.1016/j.brat.2008.02.003. Epub 2008 Feb 14. PMID 18359005
- [Result] Page AC, Hooke GR, Morrison DL. Psychometric properties of the Depression Anxiety Stress Scales (DASS) in depressed clinical samples. Br J Clin Psychol. 2007 Sep;46(Pt 3):283-97. doi: 10.1348/014466506X158996. PMID 17697478
- [Result] Radomsky, A. S., Rachman, S., Shafran, R., Coughtrey, A. E., & Barber, K. C. (2014). The nature and assessment of mental contamination: A psychometric analysis. Journal of Obsessive-Compulsive and Related Disorders, 3(2), 181-187.
- [Result] Reas DL, Grilo CM, Masheb RM. Reliability of the Eating Disorder Examination-Questionnaire in patients with binge eating disorder. Behav Res Ther. 2006 Jan;44(1):43-51. doi: 10.1016/j.brat.2005.01.004. PMID 16301013
- [Result] Schmitt DP, Allik J. Simultaneous administration of the Rosenberg Self-Esteem Scale in 53 nations: exploring the universal and culture-specific features of global self-esteem. J Pers Soc Psychol. 2005 Oct;89(4):623-42. doi: 10.1037/0022-3514.89.4.623. PMID 16287423
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Derived] Kothari R, Barker C, Pistrang N, Rozental A, Egan S, Wade T, Allcott-Watson H, Andersson G, Shafran R. A randomised controlled trial of guided internet-based cognitive behavioural therapy for perfectionism: Effects on psychopathology and transdiagnostic processes. J Behav Ther Exp Psychiatry. 2019 Sep;64:113-122. doi: 10.1016/j.jbtep.2019.03.007. Epub 2019 Mar 30. PMID 30981162
- [Derived] Shafran R, Wade TD, Egan SJ, Kothari R, Allcott-Watson H, Carlbring P, Rozental A, Andersson G. Is the devil in the detail? A randomised controlled trial of guided internet-based CBT for perfectionism. Behav Res Ther. 2017 Aug;95:99-106. doi: 10.1016/j.brat.2017.05.014. Epub 2017 May 26. PMID 28618299
- [Derived] Kothari R, Egan S, Wade T, Andersson G, Shafran R. Overcoming Perfectionism: Protocol of a Randomized Controlled Trial of an Internet-Based Guided Self-Help Cognitive Behavioral Therapy Intervention. JMIR Res Protoc. 2016 Nov 11;5(4):e215. doi: 10.2196/resprot.6378. PMID 27836815